CLINICAL TRIAL: NCT03802188
Title: Hydroxychloroquine Exposure in Systemic Lupus Erythematosus (SLE)
Brief Title: Hydroxychloroquine in Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Laval University (Other); University of British Columbia (Other); University of Calgary (Other); Dalhousie University (Other); University of Manitoba (Other); University of Toronto (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Dr. Sasha Bernatsky, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: MP-37-2019-4340
Record Dates: First submitted 2018-12-06; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Retinal toxicity
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLE Cohort: Investigators will use existing data collected on adult SLE patients enrolled into respective study cohorts from participating centers.
- Qualitative group: For the interviews, patients with SLE who are currently or have taken Hydroxychloroquine will be recruited from rheumatology clinics in Calgary and Montreal to participate in an interview and/or participate in a brief survey.

SUMMARY:
A Systemic lupus erythematosus, SLE is disease in which immune system is over-active causing inflammation in joints skin or any organ system. There are many areas where better approaches in SLE could improve outcomes. One example relates to hydroxychloroquine (HCQ) key drug which can reduce risk of serious disease flares. There are increasing concerns about eye damage main side effect with long-term use of HCQ. At present investigators cannot precisely predict which SLE patient is most likely to flare once HCQ is tapered. It is not clear what drives risk of eye damage. Investigators' study will fill these knowledge gaps. Investigators' hypothesis is that baseline demographic and clinical factors are associated with risk of SLE flare after HCQ taper/discontinuation and with risk of retinal toxicity in all HCQ exposed patients. Research will link and analyze data on 3700 SLE patients across Canada.

DETAILED DESCRIPTION:
B OBJECTIVES B1 To evaluate in SLE patients who lower but do not discontinue HCQ factors associated with flare (significant increase in disease activity, augmentation of therapy or hospitalization for SLE).

B2 To determine in SLE patients who discontinue HCQ factors associated with flare (significant increase in disease activity, therapy augmentation or hospitalization for SLE).

B3 To evaluate temporal relationship between HCQ use and retinal toxicity in SLE patients and how this may be associated with demographic and clinical factors.

B4 To assess SLE patient preferences for HCQ therapy and how preferences are associated with demographic and clinical factors.

B5 To evaluate temporal relationship between antimalarial use and other forms of toxicity in SLE patients and how this may be associated with demographic and clinical factors.

Team members have prospectively followed cohorts > 3700 adult SLE patients (90% HCQ exposed) with collected and harmonized data on demographics and clinical factors. Team members (Bernatsky Abrahamowicz Fortin Hazlewood) are founding members of CAN-AIM CIHR-funded Drug Safety and Effectiveness Network team.

Members have history of working with patients as research partners (Bartlett Li Bernatsky Fortin Hazlewood). Investigators' ties to stakeholders including patient research partners and Lupus Canada facilitates knowledge translation.

METHODS C1 Cohorts: Investigators will use existing data on adult SLE patients enrolled into study cohorts in Montreal Quebec Halifax Winnipeg Calgary and Toronto.

Investigators are members of national (Canadian Network for Improved Outcomes in SLE CaNIOS) and/or international (Systemic Lupus International Collaborating Clinics SLICC) research networks. CaNIOS and SLICC have worked decades on harmonized approach to prospectively-collected. Cohorts enroll unselected patients when they present to clinic. At annual assessments data are collected on drugs disease activity organ damage etc C2.1 Patient selection for Objective 1: At baseline and follow up visits records are made of patient HCQ doses. Starting with first visit with HCQ exposure investigators will determine how many patients are recorded as receiving lower dose or discontinuing HCQ at follow-up visit. Patients identified as having lowered HCQ dose will form sub-cohort for time-to-event (survival) analyses. Investigators will evaluate only first-ever lowering of HCQ. Analysis will evaluate patients from time zero (annual visit at which lower HCQ dose was recorded) to assess combined outcome of earliest of a) increase in SLEDAI-2K of at least 4 points and/or b) hospitalization for SLE and/or c) augmented SLE therapy defined as increase in HCQ or new start or increase in corticosteroids or other immunosuppressant. In addition to accepted minimal clinically significant SLEDAI-2K change investigators include drug changes and SLE-related hospitalizations.

Patients studied in Objective 1 will be right censored if HCQ is discontinued completely; these will enter into analyses for Objective 2. Otherwise patients will be followed until outcome of interest or end of study.

C2.3 Subject selection for Objective 2 Analyses will be similarly conducted but time zero will begin when individual discontinues HCQ. Objective 1 and 2 analyses conducted separately; patients who have HCQ dose lowered but then discontinued will be in analyses for Objective 1 up to point of discontinuation then patients will be right censored for Objective 1. Subjects are able to contribute data (from the point of HCQ discontinuation) to analyses for Objective 2. Patient can contribute to analyses for one or both objectives and contributing to Objective 3. If not right-censored patients will be followed until outcome of interest or end of study.

C2.3 Subject selection for Objective 3 Outcome is retinal toxicity assessed in HCQ-exposed patients from time of first visit with HCQ exposure up to time of retinal toxicity documentation or end of study for patients without outcome. Exposure to CQ (relatively uncommon drug exposure) is also risk factor for retinal toxicity but essentially patients exposed to CQ will have prior exposure to HCQ.

C3 Demographic and clinical factors C3.1 Variables assessed include sex age at SLE onset and race/ethnicity. Analyses adjusted for education as education can alter adherence.

C3.2 Clinical factors for multivariable analyses include smoking BMI baseline disease activity malignancy data and renal damage. Baseline refers to time zero. Renal damage is captured with SLICC Damage Index measuring accumulated damage. Baseline disease activity measured by internationally used SLEDAI-2K reliable validated widely used global score index.Investigators will model time-varying drug exposures with step-up approach initially with baseline use ie current, recent, ever or total past dose. Investigators use sophisticated and novel weighted cumulative dose modelling to flexibly represent exposures accumulated by individual subjects up to given time-point corresponding to each risk set for time-to-event analyses. In multivariable analyses approach will allow investigators to explore how risk of retinal toxicity may depend on details of past HCQ exposure including not only total cumulative dose but temporal pattern of doses at various time in past with differential weights for early versus later exposures.

C4 Outcome assessment: SLEDAI-2K and drugs are recorded. SLICC Damage Index has item for retinal damage and updated yearly.

C5 Model development: Investigators will perform multivariable time-to-event analyses in patients who lower or discontinue HCQ. Data for outcomes are available longitudinally at annual visit with actual dates only available for addition/increase in corticosteroid or SLE hospitalization. For other outcomes investigators will deal with interval-censored data familiar issue in pharmacoepidemiology.

Models include baseline demographics education BMI SLE duration SLEDAI-2K renal damage and medications. Simplistic survival analyses often assume linear effects of continuous covariates and impose conventional proportional hazards (PH) assumptions; investigators know that prognostic factors may have time-dependent and/or nonlinear effects that violate assumptions. Investigators will account for this. Methods account for possible changes in hazard ratio over time (violation of the PH) and allow estimation of relative risks (hazard ratios) and actual probabilities of event of interest occurring.

Similar approach will be used for Objective 3 in time-to-event analyses of retinal toxicity in patients exposed to HCQ.

Competing risks occur when subjects can experience one or more events that may compete with outcome of interest and hinder observation of event of interest or modify chances for event to occur. In sensitivity analyses investigators use competing risks models to simultaneously estimate associations between HCQ exposures and hazards of competing event.

D POWER/SAMPLE CALCULATIONS D1 Power calculations for multivariate models Combined cohorts include over 3300 patients have exposed to HCQ. Patients have had lowering of dose 45% or discontinuation of HCQ during their follow-up. Power calculations are based on available data suggesting that 45%-60% of SLE patients may flare over ten years of follow-up.

For baseline SLEDAI-2K assuming 35% of patients score less than 3 investigators would have 90% power to detect unadjusted HR of 1.30 and adjusted HR of 1.37 for variable. Assuming 20% of patients have renal damage investigators will have 90% power to detect an unadjusted HR of 1.37 and an adjusted HR of 1.45 for variable.

E KNOWLEDGE TRANSLATION activities are informed by history of partnerships between investigators and knowledge-users directed by Dr. Linda Li Canada Research Chair in Patient-Oriented KT and Director of Knowledge Translation Research Program at UBC's Arthritis Research Centre of Canada.

E1 Integrated KT Proposal developed in consultation patients from Lupus Canada patients Canadian Alliance of Patients with Arthritis (CAPA) and Singer Family Fund for Lupus Research. Wendy Singer (providing expertise health information dissemination and provides insight of SLE patient who has been affected by HCQ-induced retinal toxicity) will assist with educational tool developments. Co-PI Dr. Bartlett has over decade of work with patient partners through OMERACT (Outcome Measures in Rheumatology) and other organizations to help disseminate findings patient communities.

E2 Dissemination via MyLupusGuide: Data on HCQ from current study will be incorporated into MyLupusGuide web-based patient-centred health-management tool developed by Dr. Fortin in partnership with Jack Digital Productions CaNIOS Lupus Canada. Development validation/dissemination of current version funded by CIHR operating and dissemination grants.

E3 Clinicians and professional groups: Dr. Bernatsky is member of CRA Therapeutics Committee which advises CRA on policies related to drug use for rheumatic diseases. Group monitors information about adverse events related to drugs used in rheumatology including HCQ. Investigators submit abstracts to scientific meetings (American College of Rheumatology, European League Against Rheumatism, CRA meeting). Investigators will seek feedback on feasibility/approaches to integrate MyLupusGuide as gold standard for patient education tool concerning HCQ.

E4 Informing future guidelines: Team member Dr. S. Keeling has already produced Canadian SLE care guidelines (funded by the CIHR and endorsed by the CRA and CaNIOS) . In 2019, again mandated by these groups, Dr. Keeling will spearhead guidelines for SLE therapies.

E5 Health agency stakeholders: Investigators have connections Drug Safety and Effectiveness Network (DSEN) Health Canada's Marketed Health Product Directorate and Canadian Agency for Drugs and Technologies in Health (CADTH). Drs. Abrahamowicz and Bernatsky are co-leads DSEN-funded team.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or over
* Must be diagnosed with Systemic Lupus Erythematosus (SLE)
* Must be exposed to hydroxychloroquine
* Must be enrolled at participating sites

Exclusion Criteria:

* Under 18 years of age
* Not diagnosed with SLE
* Not exposed to hydroxychloroquine
* Not enrolled at participating sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will use existing data collected on adult SLE patients who have been consecutively enrolled into the respective study cohorts of the participating researchers in Montreal , Quebec City, Halifax, Winnipeg, Calgary, and Toronto. The total exceeds 3,300 SLE patients who have been exposed to HCQ.
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of SLE flares with decrease or discontinuation of HCQ | Through study completion, an average of 1 year
  In patients exposed to HCQ, presence or absence of SLE flare will be measure with SLEDAI-2K. The SLEDAI-2K is a reliable, validated, widely used global score index, consisting of 24 weighted clinical and laboratory variables of nine organ systems. The scores of descriptors range from 1 to 8, and the total score of the SLEDAI-2K is the sum of all 24 descriptor scores. An increase of 4 points or more has been validated as indicating a clinically significant increase in SLE disease activity.

SECONDARY OUTCOMES:
Proportion of participants hospitalized with decrease or discontinuation of HCQ | Through study completion, an average of 1 year
  In patients exposed to HCQ, presence or absence of hospitalization in cohort data will be measured in relation to HCQ dosage.
Proportion of SLE flares relative to augmented SLE therapy | Through study completion, an average of 1 year
  Comparison of flares in SLE patients measured with SLEDAI-2K and augmented SLE therapy defined as an increase in HCQ or a new start or increase in corticosteroids (i.e. prednisone, methylprednisolone) or other immunosuppressant (azathioprine, mycophenolate, methotrexate, cyclophosphamide, belimumab, rituximab, chloroquine).
Correlation of retinal toxicity and exposure to HCQ and retinal toxicity | Through study completion, an average of 1 year
  Renal damage is captured with the SLICC Damage Index, measuring accumulated damage since SLE onset. This validated index captures irreversible change in an organ or system (that has been present for at least 6 months). The renal item scores 1 for sustained heavy proteinuria, 2 for reduced glomerular filtration rate, and 3 for end-stage renal failure.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Bernatsky, MD/PhD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keeling SO, Alabdurubalnabi Z, Avina-Zubieta A, Barr S, Bergeron L, Bernatsky S, Bourre-Tessier J, Clarke A, Baril-Dionne A, Dutz J, Ensworth S, Fifi-Mah A, Fortin PR, Gladman DD, Haaland D, Hanly JG, Hiraki LT, Hussein S, Legault K, Levy D, Lim L, Matsos M, McDonald EG, Medina-Rosas J, Pardo Pardi J, Peschken C, Pineau C, Pope J, Rader T, Reynolds J, Silverman E, Tselios K, Suitner M, Urowitz M, Touma Z, Vinet E, Santesso N. Canadian Rheumatology Association Recommendations for the Assessment and Monitoring of Systemic Lupus Erythematosus. J Rheumatol. 2018 Oct;45(10):1426-1439. doi: 10.3899/jrheum.171459. Epub 2018 Sep 1. PMID 30173152
- [Background] Jonsen A, Clarke AE, Joseph L, Belisle P, Bernatsky S, Nived O, Bengtsson AA, Sturfelt G, Pineau CA. Association of the Charlson comorbidity index with mortality in systemic lupus erythematosus. Arthritis Care Res (Hoboken). 2011 Sep;63(9):1233-7. doi: 10.1002/acr.20506. PMID 21618451
- [Background] Akhavan PS, Su J, Lou W, Gladman DD, Urowitz MB, Fortin PR. The early protective effect of hydroxychloroquine on the risk of cumulative damage in patients with systemic lupus erythematosus. J Rheumatol. 2013 Jun;40(6):831-41. doi: 10.3899/jrheum.120572. Epub 2013 Apr 15. PMID 23588942
- [Background] Levy DM, Peschken CA, Tucker LB, Chedeville G, Huber AM, Pope JE; Canadian Network for Improved Outcomes in SLE (CaNIOS) 1000 Faces Investigators; Silverman ED. Association of health-related quality of life in childhood-onset systemic lupus erythematosus with ethnicity: results from a multiethnic multicenter Canadian cohort. Arthritis Care Res (Hoboken). 2014 Dec;66(12):1767-74. doi: 10.1002/acr.22363. PMID 24821613
- [Background] Aghdassi E, Zhang W, St-Pierre Y, Clarke AE, Morrison S, Peeva V, Landolt-Marticorena C, Su J, Reich H, Scholey J, Herzenberg A, Pope JE, Peschken C; LuNNET CaNIOS Investigators; Wither JE, Fortin PR. Healthcare cost and loss of productivity in a Canadian population of patients with and without lupus nephritis. J Rheumatol. 2011 Apr;38(4):658-66. doi: 10.3899/jrheum.100482. Epub 2010 Dec 15. PMID 21159829
- [Background] Peschken CA, Katz SJ, Silverman E, Pope JE, Fortin PR, Pineau C, Smith CD, Arbillaga HO, Gladman DD, Urowitz M, Zummer M, Clarke A, Bernatsky S, Hudson M; Canadian Network for Improved Outcomes in Systemic Lupus Erythematosus (CaNIOS). The 1000 Canadian faces of lupus: determinants of disease outcome in a large multiethnic cohort. J Rheumatol. 2009 Jun;36(6):1200-8. doi: 10.3899/jrheum.080912. Epub 2009 Apr 15. PMID 19369456
- [Background] Bruce IN, O'Keeffe AG, Farewell V, Hanly JG, Manzi S, Su L, Gladman DD, Bae SC, Sanchez-Guerrero J, Romero-Diaz J, Gordon C, Wallace DJ, Clarke AE, Bernatsky S, Ginzler EM, Isenberg DA, Rahman A, Merrill JT, Alarcon GS, Fessler BJ, Fortin PR, Petri M, Steinsson K, Dooley MA, Khamashta MA, Ramsey-Goldman R, Zoma AA, Sturfelt GK, Nived O, Aranow C, Mackay M, Ramos-Casals M, van Vollenhoven RF, Kalunian KC, Ruiz-Irastorza G, Lim S, Kamen DL, Peschken CA, Inanc M, Urowitz MB. Factors associated with damage accrual in patients with systemic lupus erythematosus: results from the Systemic Lupus International Collaborating Clinics (SLICC) Inception Cohort. Ann Rheum Dis. 2015 Sep;74(9):1706-13. doi: 10.1136/annrheumdis-2013-205171. Epub 2014 May 16. PMID 24834926
- [Background] Lee J, Dhillon N, Pope J. All-cause hospitalizations in systemic lupus erythematosus from a large Canadian referral centre. Rheumatology (Oxford). 2013 May;52(5):905-9. doi: 10.1093/rheumatology/kes391. Epub 2013 Jan 9. PMID 23307831
- [Background] Garcia-Gonzalez A, Richardson M, Garcia Popa-Lisseanu M, Cox V, Kallen MA, Janssen N, Ng B, Marcus DM, Reveille JD, Suarez-Almazor ME. Treatment adherence in patients with rheumatoid arthritis and systemic lupus erythematosus. Clin Rheumatol. 2008 Jul;27(7):883-9. doi: 10.1007/s10067-007-0816-6. Epub 2008 Jan 8. PMID 18185905
- [Background] Koneru S, Kocharla L, Higgins GC, Ware A, Passo MH, Farhey YD, Mongey AB, Graham TB, Houk JL, Brunner HI. Adherence to medications in systemic lupus erythematosus. J Clin Rheumatol. 2008 Aug;14(4):195-201. doi: 10.1097/RHU.0b013e31817a242a. PMID 18636020
- [Background] Mehat P, Atiquzzaman M, Esdaile JM, AviNa-Zubieta A, De Vera MA. Medication Nonadherence in Systemic Lupus Erythematosus: A Systematic Review. Arthritis Care Res (Hoboken). 2017 Nov;69(11):1706-1713. doi: 10.1002/acr.23191. Epub 2017 Sep 21. PMID 28086003
- [Background] Leroux G, Costedoat-Chalumeau N, Hulot JS, Amoura Z, Frances C, Aymard G, Lechat P, Piette JC. Relationship between blood hydroxychloroquine and desethylchloroquine concentrations and cigarette smoking in treated patients with connective tissue diseases. Ann Rheum Dis. 2007 Nov;66(11):1547-8. doi: 10.1136/ard.2007.072587. No abstract available. PMID 17934086
- [Background] Dixon WG, Abrahamowicz M, Beauchamp ME, Ray DW, Bernatsky S, Suissa S, Sylvestre MP. Immediate and delayed impact of oral glucocorticoid therapy on risk of serious infection in older patients with rheumatoid arthritis: a nested case-control analysis. Ann Rheum Dis. 2012 Jul;71(7):1128-33. doi: 10.1136/annrheumdis-2011-200702. Epub 2012 Jan 12. PMID 22241902
- [Background] Widdifield J, Moura CS, Wang Y, Abrahamowicz M, Paterson JM, Huang A, Beauchamp ME, Boire G, Fortin PR, Bessette L, Bombardier C, Hanly JG, Feldman D, Bernatsky S; CAnadian Network for Advanced Interdisciplinary Methods for comparative effectiveness research (CAN-AIM). The Longterm Effect of Early Intensive Treatment of Seniors with Rheumatoid Arthritis: A Comparison of 2 Population-based Cohort Studies on Time to Joint Replacement Surgery. J Rheumatol. 2016 May;43(5):861-8. doi: 10.3899/jrheum.151156. Epub 2016 Feb 15. PMID 26879353
- [Background] Moura CS, Abrahamowicz M, Beauchamp ME, Lacaille D, Wang Y, Boire G, Fortin PR, Bessette L, Bombardier C, Widdifield J, Hanly JG, Feldman D, Maksymowych W, Peschken C, Barnabe C, Edworthy S, Bernatsky S; CAN-AIM. Early medication use in new-onset rheumatoid arthritis may delay joint replacement: results of a large population-based study. Arthritis Res Ther. 2015 Aug 3;17(1):197. doi: 10.1186/s13075-015-0713-3. PMID 26235697
- [Background] Sylvestre MP, Abrahamowicz M. Flexible modeling of the cumulative effects of time-dependent exposures on the hazard. Stat Med. 2009 Nov 30;28(27):3437-53. doi: 10.1002/sim.3701. PMID 19708037
- [Background] Marmor MF, Carr RE, Easterbrook M, Farjo AA, Mieler WF; American Academy of Ophthalmology. Recommendations on screening for chloroquine and hydroxychloroquine retinopathy: a report by the American Academy of Ophthalmology. Ophthalmology. 2002 Jul;109(7):1377-82. doi: 10.1016/s0161-6420(02)01168-5. No abstract available. PMID 12093666
- [Background] Sun X, Li X, Chen C, Song Y. A review of statistical issues with progression-free survival as an interval-censored time-to-event endpoint. J Biopharm Stat. 2013;23(5):986-1003. doi: 10.1080/10543406.2013.813524. PMID 23957511
- [Background] Wynant W, Abrahamowicz M. Flexible estimation of survival curves conditional on non-linear and time-dependent predictor effects. Stat Med. 2016 Feb 20;35(4):553-65. doi: 10.1002/sim.6740. Epub 2015 Nov 6. PMID 26542758
- [Background] Wynant W, Abrahamowicz M. Impact of the model-building strategy on inference about nonlinear and time-dependent covariate effects in survival analysis. Stat Med. 2014 Aug 30;33(19):3318-37. doi: 10.1002/sim.6178. Epub 2014 Apr 22. PMID 24757068
- [Background] Reed Johnson F, Lancsar E, Marshall D, Kilambi V, Muhlbacher A, Regier DA, Bresnahan BW, Kanninen B, Bridges JF. Constructing experimental designs for discrete-choice experiments: report of the ISPOR Conjoint Analysis Experimental Design Good Research Practices Task Force. Value Health. 2013 Jan-Feb;16(1):3-13. doi: 10.1016/j.jval.2012.08.2223. PMID 23337210
- [Background] Black N, Burke L, Forrest CB, Sieberer UH, Ahmed S, Valderas JM, Bartlett SJ, Alonso J. Patient-reported outcomes: pathways to better health, better services, and better societies. Qual Life Res. 2016 May;25(5):1103-12. doi: 10.1007/s11136-015-1168-3. Epub 2015 Nov 13. PMID 26563251
- [Background] Neville C, DaCosta D, Rochon M, Eng D, Fortin PR. Toward the development of a lupus interactive navigator to facilitate patients and their health care providers in the management of lupus: results of web-based surveys. JMIR Res Protoc. 2014 Dec 22;3(4):e65. doi: 10.2196/resprot.3349. PMID 25533760
- [Background] Bernatsky S, Peschken C, Fortin PR, Pineau CA, Urowitz MB, Gladman DD, Pope JE, Hudson M, Zummer M, Smith CD, Arbillaga HO, Clarke AE; Canadian Network for Improved Outcomes in Systemic Lupus Erythematosus (CaNIOS). Medication use in systemic lupus erythematosus. J Rheumatol. 2011 Feb;38(2):271-4. doi: 10.3899/jrheum.100414. Epub 2010 Nov 15. PMID 21078722
- [Background] Clarke AE, Urowitz MB, Monga N, Hanly JG. Costs associated with severe and nonsevere systemic lupus erythematosus in Canada. Arthritis Care Res (Hoboken). 2015 Mar;67(3):431-6. doi: 10.1002/acr.22452. PMID 25185936
- [Background] Mahler M, Parker T, Peebles CL, Andrade LE, Swart A, Carbone Y, Ferguson DJ, Villalta D, Bizzaro N, Hanly JG, Fritzler MJ. Anti-DFS70/LEDGF antibodies are more prevalent in healthy individuals compared to patients with systemic autoimmune rheumatic diseases. J Rheumatol. 2012 Nov;39(11):2104-10. doi: 10.3899/jrheum.120598. Epub 2012 Sep 1. PMID 22942262
- [Background] Furst DE, Clarke A, Fernandes AW, Bancroft T, Gajria K, Greth W, Iorga SR. Resource utilization and direct medical costs in adult systemic lupus erythematosus patients from a commercially insured population. Lupus. 2013 Mar;22(3):268-78. doi: 10.1177/0961203312474087. Epub 2013 Jan 22. PMID 23340996
- [Background] Isenberg DA, Gladman D. The Systemic Lupus International Collaborating Clinics Group--origins and outcomes. Lupus. 2001;10(5):375-7. doi: 10.1191/096120301676101377. No abstract available. PMID 11403271
- [Background] Isenberg DA, Ramsey-Goldman R, Gladman D, Hanly JG. The Systemic Lupus International Collaborating Clinics (SLICC) group - it was 20 years ago today. Lupus. 2011 Nov;20(13):1426-32. doi: 10.1177/0961203311421501. PMID 22095889
- [Background] Lee J, Peschken CA, Muangchan C, Silverman E, Pineau C, Smith CD, Arbillaga H, Zummer M, Clarke A, Bernatsky S, Hudson M, Hitchon C, Fortin PR, Pope JE. The frequency of and associations with hospitalization secondary to lupus flares from the 1000 Faces of Lupus Canadian cohort. Lupus. 2013 Nov;22(13):1341-8. doi: 10.1177/0961203313505689. Epub 2013 Sep 18. PMID 24048215
- [Background] Bernatsky S, Ramsey-Goldman R, Labrecque J, Joseph L, Boivin JF, Petri M, Zoma A, Manzi S, Urowitz MB, Gladman D, Fortin PR, Ginzler E, Yelin E, Bae SC, Wallace DJ, Edworthy S, Jacobsen S, Gordon C, Dooley MA, Peschken CA, Hanly JG, Alarcon GS, Nived O, Ruiz-Irastorza G, Isenberg D, Rahman A, Witte T, Aranow C, Kamen DL, Steinsson K, Askanase A, Barr S, Criswell LA, Sturfelt G, Patel NM, Senecal JL, Zummer M, Pope JE, Ensworth S, El-Gabalawy H, McCarthy T, Dreyer L, Sibley J, St Pierre Y, Clarke AE. Cancer risk in systemic lupus: an updated international multi-centre cohort study. J Autoimmun. 2013 May;42:130-5. doi: 10.1016/j.jaut.2012.12.009. Epub 2013 Feb 12. PMID 23410586
- [Background] Bernatsky S, Ramsey-Goldman R, Joseph L, Boivin JF, Costenbader KH, Urowitz MB, Gladman DD, Fortin PR, Nived O, Petri MA, Jacobsen S, Manzi S, Ginzler EM, Isenberg D, Rahman A, Gordon C, Ruiz-Irastorza G, Yelin E, Bae SC, Wallace DJ, Peschken CA, Dooley MA, Edworthy SM, Aranow C, Kamen DL, Romero-Diaz J, Askanase A, Witte T, Barr SG, Criswell LA, Sturfelt GK, Blanco I, Feldman CH, Dreyer L, Patel NM, St Pierre Y, Clarke AE. Lymphoma risk in systemic lupus: effects of disease activity versus treatment. Ann Rheum Dis. 2014 Jan;73(1):138-42. doi: 10.1136/annrheumdis-2012-202099. Epub 2013 Jan 8. PMID 23303389
- [Background] Bernatsky S, Clarke A, Gladman DD, Urowitz M, Fortin PR, Barr SG, Senecal JL, Zummer M, Edworthy S, Sibley J, Pope J, Ensworth S, Ramsey-Goldman R, Hanly JG. Mortality related to cerebrovascular disease in systemic lupus erythematosus. Lupus. 2006;15(12):835-9. doi: 10.1177/0961203306073133. PMID 17211987
- [Background] Bernatsky S, Boivin JF, Joseph L, Manzi S, Ginzler E, Gladman DD, Urowitz M, Fortin PR, Petri M, Barr S, Gordon C, Bae SC, Isenberg D, Zoma A, Aranow C, Dooley MA, Nived O, Sturfelt G, Steinsson K, Alarcon G, Senecal JL, Zummer M, Hanly J, Ensworth S, Pope J, Edworthy S, Rahman A, Sibley J, El-Gabalawy H, McCarthy T, St Pierre Y, Clarke A, Ramsey-Goldman R. Mortality in systemic lupus erythematosus. Arthritis Rheum. 2006 Aug;54(8):2550-7. doi: 10.1002/art.21955. PMID 16868977
- [Background] Lu M, Bernatsky S, Ramsey-Goldman R, Petri M, Manzi S, Urowitz MB, Gladman D, Fortin PR, Ginzler EM, Yelin E, Bae SC, Wallace DJ, Jacobsen S, Dooley MA, Peschken CA, Alarcon GS, Nived O, Gottesman L, Criswell LA, Sturfelt G, Dreyer L, Lee JL, Clarke AE. Non-lymphoma hematological malignancies in systemic lupus erythematosus. Oncology. 2013;85(4):235-40. doi: 10.1159/000350165. Epub 2013 Oct 2. PMID 24107608
- [Background] Steiner JF, Koepsell TD, Fihn SD, Inui TS. A general method of compliance assessment using centralized pharmacy records. Description and validation. Med Care. 1988 Aug;26(8):814-23. doi: 10.1097/00005650-198808000-00007. PMID 3398608
- [Result] Bernatsky S, Joseph L, Pineau CA, Tamblyn R, Feldman DE, Clarke AE. A population-based assessment of systemic lupus erythematosus incidence and prevalence--results and implications of using administrative data for epidemiological studies. Rheumatology (Oxford). 2007 Dec;46(12):1814-8. doi: 10.1093/rheumatology/kem233. PMID 18032538
- [Result] Canadian Hydroxychloroquine Study Group. A randomized study of the effect of withdrawing hydroxychloroquine sulfate in systemic lupus erythematosus. N Engl J Med. 1991 Jan 17;324(3):150-4. doi: 10.1056/NEJM199101173240303. PMID 1984192
- [Result] Tsakonas E, Joseph L, Esdaile JM, Choquette D, Senecal JL, Cividino A, Danoff D, Osterland CK, Yeadon C, Smith CD. A long-term study of hydroxychloroquine withdrawal on exacerbations in systemic lupus erythematosus. The Canadian Hydroxychloroquine Study Group. Lupus. 1998;7(2):80-5. doi: 10.1191/096120398678919778. PMID 9541091
- [Result] Waldron N, Brown S, Hewlett S, Elliott B, McHugh N, McCabe C. 'It's more scary not to know': a qualitative study exploring the information needs of patients with systemic lupus erythematosus at the time of diagnosis. Musculoskeletal Care. 2011 Dec;9(4):228-38. doi: 10.1002/msc.221. Epub 2011 Oct 13. PMID 21993962
- [Result] Telek HH, Yesilirmak N, Sungur G, Ozdemir Y, Yesil NK, Ornek F. Retinal toxicity related to hydroxychloroquine in patients with systemic lupus erythematosus and rheumatoid arthritis. Doc Ophthalmol. 2017 Dec;135(3):187-194. doi: 10.1007/s10633-017-9607-9. Epub 2017 Aug 29. PMID 28852896
- [Result] Gladman D, Ginzler E, Goldsmith C, Fortin P, Liang M, Urowitz M, Bacon P, Bombardieri S, Hanly J, Hay E, Isenberg D, Jones J, Kalunian K, Maddison P, Nived O, Petri M, Richter M, Sanchez-Guerrero J, Snaith M, Sturfelt G, Symmons D, Zoma A. The development and initial validation of the Systemic Lupus International Collaborating Clinics/American College of Rheumatology damage index for systemic lupus erythematosus. Arthritis Rheum. 1996 Mar;39(3):363-9. doi: 10.1002/art.1780390303. PMID 8607884
- [Result] Yee CS, Farewell VT, Isenberg DA, Griffiths B, Teh LS, Bruce IN, Ahmad Y, Rahman A, Prabu A, Akil M, McHugh N, Edwards C, D'Cruz D, Khamashta MA, Gordon C. The use of Systemic Lupus Erythematosus Disease Activity Index-2000 to define active disease and minimal clinically meaningful change based on data from a large cohort of systemic lupus erythematosus patients. Rheumatology (Oxford). 2011 May;50(5):982-8. doi: 10.1093/rheumatology/keq376. Epub 2011 Jan 18. PMID 21245073
- [Result] Ward MM, Marx AS, Barry NN. Comparison of the validity and sensitivity to change of 5 activity indices in systemic lupus erythematosus. J Rheumatol. 2000 Mar;27(3):664-70. PMID 10743805
- [Result] Satagopan JM, Ben-Porat L, Berwick M, Robson M, Kutler D, Auerbach AD. A note on competing risks in survival data analysis. Br J Cancer. 2004 Oct 4;91(7):1229-35. doi: 10.1038/sj.bjc.6602102. PMID 15305188
- [Result] Hazlewood GS, Bombardier C, Tomlinson G, Thorne C, Bykerk VP, Thompson A, Tin D, Marshall DA. Treatment preferences of patients with early rheumatoid arthritis: a discrete-choice experiment. Rheumatology (Oxford). 2016 Nov;55(11):1959-1968. doi: 10.1093/rheumatology/kew280. Epub 2016 Jul 31. PMID 27477807
- [Result] Petri M, Genovese M, Engle E, Hochberg M. Definition, incidence, and clinical description of flare in systemic lupus erythematosus. A prospective cohort study. Arthritis Rheum. 1991 Aug;34(8):937-44. doi: 10.1002/art.1780340802. PMID 1859487
- [Result] Hoaglin DC, Hawkins N, Jansen JP, Scott DA, Itzler R, Cappelleri JC, Boersma C, Thompson D, Larholt KM, Diaz M, Barrett A. Conducting indirect-treatment-comparison and network-meta-analysis studies: report of the ISPOR Task Force on Indirect Treatment Comparisons Good Research Practices: part 2. Value Health. 2011 Jun;14(4):429-37. doi: 10.1016/j.jval.2011.01.011. PMID 21669367
- [Result] Haase KR, Loiselle CG. Oncology team members' perceptions of a virtual navigation tool for cancer patients. Int J Med Inform. 2012 Jun;81(6):395-403. doi: 10.1016/j.ijmedinf.2011.11.001. Epub 2012 Jan 13. PMID 22244817
- [Result] Loiselle CG, Peters O, Haase KR, Girouard L, Korner A, Wiljer D, Fitch M. Virtual navigation in colorectal cancer and melanoma: an exploration of patients' views. Support Care Cancer. 2013 Aug;21(8):2289-96. doi: 10.1007/s00520-013-1771-1. Epub 2013 Mar 22. PMID 23519565
- [Result] Neville C, Da Costa D, Rochon M, Peschken CA, Pineau CA, Bernatsky S, Keeling S, Avina-Zubieta A, Lye E, Eng D, Fortin PR. Development of the Lupus Interactive Navigator as an Empowering Web-Based eHealth Tool to Facilitate Lupus Management: Users Perspectives on Usability and Acceptability. JMIR Res Protoc. 2016 May 30;5(2):e44. doi: 10.2196/resprot.4219. PMID 27240666
- [Result] Moss KE, Ioannou Y, Sultan SM, Haq I, Isenberg DA. Outcome of a cohort of 300 patients with systemic lupus erythematosus attending a dedicated clinic for over two decades. Ann Rheum Dis. 2002 May;61(5):409-13. doi: 10.1136/ard.61.5.409. PMID 11959764
- [Result] Clowse ME, Magder L, Witter F, Petri M. Hydroxychloroquine in lupus pregnancy. Arthritis Rheum. 2006 Nov;54(11):3640-7. doi: 10.1002/art.22159. PMID 17075810
- See also: AAO Quality of Care Secretariat, Hoskins Center for Quality Eye Care Recommendations on Screening for Chloroquine and Hydroxychloroquine Retinopathy Ophthalmology — https://www.aao.org/clinical-statement/revised-recommendations-on-screening-chloroquine-h
- See also: CAnadian Network for Advanced Interdisciplinary Methods for comparative effectiveness research — http://canaim.ca/about-us
- See also: Lack of Interferon and Proinflammatory Cyto/chemokines in Serologically Active Clinically Quiescent SLE. — http://www.jrheum.org/content/42/12/2318.full.pdf
- See also: Racial and Ethnic Categories and Definitions — https://grants.nih.gov/grants/guide/rfa-files/RFA-OD-19-012.html
- See also: Purposeful sampling for qualitative data collection and analysis in mixed method implementation research. Administration and policy in mental health — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4012002/
- See also: Patient Reported Outcomes in Rheumatic Diseases, Rheumatic Disease Clinics of North America — https://mapigroup.com/pro_newsletter/patient-reported-outcomes-in-rheumatic-diseases-an-issue-of-rheumatic-disease-clinics-of-north-america-1st-edition/